CLINICAL TRIAL: NCT05409248
Title: Cognitive Stimulation Intervention Program for Cancer Survivors and Its Benefit on Cognitive Performance and Quality of Life
Brief Title: Cognitive Stimulation and Chemobrain. An Innovative Intervention for Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Antonio de Nebrija (Other)
Collaborators: Hospital de la Ribera (Other)
Responsible Party: Principal Investigator, Jon Andoni Duñabeitia, Director, Universidad Antonio de Nebrija
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CSCS
Record Dates: First submitted 2021-10-14; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Breast Cancer; Cognitive Decline
Keywords: Breast cancer; Cancer survivors; Chemobrain; Cognitive stimulation; Online intervention
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction; Chemotherapy-Related Cognitive Impairment

STUDY DESIGN:
Intervention Model Description: A home-based intervention will be set through the CogniFit® online platform. Participants will access remotely from home using a personal computer or smart device. The cognitive stimulation program will be held for 5 consecutive days (Monday to Friday) for 8 weeks, completing a total of 40 training sessions. Researchers will supervise the participant's performance daily and will periodically contact participants via telephone.
Who Masked: Participant, Investigator
Masking Description: The intervention platform will randomly assign participants in a 1:1 ratio to one out of two groups (control/experimental), so both participants and researchers are blinded.
  Activities presented to the experimental group will target specific cognitive domains (mainly executive functions) and will be automatically adjusted in difficulty and requirement according to each participant's performance. Thus, maximum cognitive effort is always required.
  Activities presented to the active control group will target orthogonal unrelated cognitive domains (i.e. artistic cognitive processes) and will be of constant difficulty.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Online games designed to target specific cognitive skills such as attention, perception, or inhibition). Activities' difficulty will be automatically adjusted accordingly to each participant's performance, always demanding a maximum cognitive effort.
  Interventions: Other: Personalized cognitive stimulation
- Control Group (Active Comparator): Online painting and artistic games designed not to target the specific cognitive skills at test. Activities' duration will match those of the experimental group, and its difficulty will be constant through the intervention.
  Interventions: Other: Sham cognitive stimulation

INTERVENTIONS:
Other: Personalized cognitive stimulation — Online gamified activities designed to stimulate cognitive functions (specifically executive function) will be carried out through a mobile application or web browser. Performance feedback will be shown after each activity.
  Other Names: CogniFit's personalized brain training
  Arms: Experimental Group
Other: Sham cognitive stimulation — Non-therapeutic online games based on artistic tasks designed to not train the specific cognitive abilities at test. The time of each session will match that of the experimental group. Performance feedback will be shown after each game.
  Arms: Control Group

SUMMARY:
The present study aims to establish a non-pharmacological alternative in alleviating cognitive deterioration derived from undergoing chemotherapy treatment. Thus, the effectiveness of a personalized and computerized cognitive stimulation program in breast cancer survivors is assessed.

DETAILED DESCRIPTION:
A phase I/II/III clinical trial is proposed in which the first two phases will serve to evaluate the safety of the intervention and the maximum tolerated time of computerized cognitive training per session in the absence of adverse effects. The third phase will consist of a double-blind randomized controlled trial where the effectiveness of the personalized and self-administered computerized cognitive stimulation program will be evaluated.

Phase I. Based on a dose-escalation 3+3 design, experienced fatigue or adverse effects will be measured after succeeding 15 minutes cognitive stimulation training blocks. The training dose will be set to a block before extreme fatigue or notable adverse effect has been reported by two or more participants. A trained psychologist will supervise the process.

Phase II. To evaluate the effectiveness of the intervention, 20 participants will undertake an interspersed training day and evaluation day through 15 consecutive days. In this way, a total of 8 evaluation sessions (day 1, 3, 5, 7, 9, 11, 13, and 15) and 7 cognitive stimulation sessions (day 2, 4, 6, 8, 10, 12, and 14) will be carried out. A trained psychologist will supervise every step of the process.

Phase III. An 8-week personalized and computerized cognitive stimulation program will be established, where the training time per session will be as determined on phase I. 120 participants will be randomized 1:1 ratio to an intervention or active control group. All participants will undertake a pre and post-test, with a total of 40 training sessions (Monday to Friday) during 8 weeks. Although this phase is set to be an online home-based stage, the responsible psychologist will be monitoring participants' performance and will periodically contact participants via telephone.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with breast cancer.
* Having undergone chemotherapy.
* Report objective or subjective complaints of cognitive impairment.

Exclusion Criteria:

* Metastases or brain tumors.
* Existence of a relevant medical, psychiatric, or neurological disorder.
* Significant visual or motor impairments.
* History of alcohol or drug abuse or dependence.
* Be receiving another cognitive stimulation intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since the study population is breast cancer survivors, and considering its epidemiology, investigators will restrict participants to females.
Enrollment: 120 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in mini-Mental Adjustment to Cancer Scale (mini-MAC) at Week 8 | Baseline and Week 8
  The mini-MAC is a validated 29-item self-rated questionnaire that examines five cancer-specific coping strategies: fighting spirit, helplessness, anxious preoccupation, cognitive avoidance, and fatalism. Each item is scored using a 4-point Likert scale. Higher scores on each subscale mean greater use of that strategy.
Change from Baseline in Cognitive Assessment for Chemo Fog Research (CAB-CF) at Week 8 | Baseline and Week 8
  The CAB-CF is an online neuropsychological assessment battery that evaluates a total of 23 cognitive skills, grouped into 5 cognitive domains (attention, memory, coordination, perception, and reasoning). Each cognitive skill is scored from 0 to 800. The cognitive domain score is calculated by averaging the scores of the cognitive skills that comprise it. Higher scores mean better cognitive performance.
Change from Baseline in the Functionality Assessment Instrument in Cancer Treatment - Cognitive Function (FACT-COG) at Week 8 | Baseline and Week 8
  The FACT-COG is a 37 item self-report questionnaire that assesses patients' perception of their cognitive abilities, functionality, and quality of life. Each item is scored using a 5-point Likert scale. Higher scores indicate less perceived cognitive impairment.

SECONDARY OUTCOMES:
Change from Baseline in the State-Trait Anxiety Inventory (STAI) at Week 8 | Baseline and Week 8
  The STAI is a validated self-report that assesses anxiety that measures both trait and state anxiety. Each item is scored using a 4-point Likert scale. Possible scores range from 0 (no anxiety) to 60 (severe anxiety), for each category.
Change from Baseline in the Beck Depression Inventory (BDI-II) at Week 8 | Baseline and Week 8
  The BDI-II is a validated 21-item self-report inventory designed to measure the frequency and severity of depressive symptoms. Scores range from 0 (no depressive symptoms) to 63 (severe depression).
Change from Baseline in the Brief Fatigue Inventory (BFI) at Week 8 | Baseline and Week 8
  The BFI is a 9-items instrument designed to assess the severity and impact of cancer-related fatigue. For the three items that assess fatigue severity, scores range from 0 (no fatigue) to 10 (the worst fatigue you can imagine). For the six items that assess how fatigue interferes with daily life, scores range from 0 (does not interfere) to 10 (interferes completely).
Change from Baseline in the Measuring Quality of Life | The World Health Organization - abridged version (WHOQOL-BREF) at Week 8 | Baseline and Week 8
  The WHOQOL-BREF is a 26-question questionnaire designed to measure the quality of life. It has two questions concerning the general satisfaction with health, and the remaining 24 questions are grouped in four areas: physical health, psychological health, social relations, and environment. Scores for each domain range from 0 (poor perceived quality of life) to 100 (greater perceived quality of life)
Change from Baseline in the Columbia-Suicide Severity Rating Scale (C-SSRS) at Week 8 | Baseline and Week 8
  The C-SSRS is a questionnaire designed to assess the existence of thoughts, desires or behaviors related to suicidal ideation, assessing a total of ten categories (wish to be dead; non-specific active suicidal thoughts; active suicidal ideation with any methods without intent to act; active suicidal ideation with some intent to act, without a specific plan; active suicidal Ideation with a specific plan and intent; preparatory acts or behavior; aborted attempt; interrupted attempt; actual attempt; completed suicide. The questionnaire can be administered as a self-report, with additional open-ended follow-up questions to provide more information. Scoring refers to the presence or absence of each of the 10 categories, provided by the dichotomous responses (Yes/No).

CONTACTS AND LOCATIONS:
Overall Officials: Jon A Duñabeitia, Study Director — Universidad Nebrija; Jose L Tapia, Principal Investigator — Univerisdad Nebrija
Locations (1):
- Hospital la Ribera, Alzira, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
The data protection policy of the public health system of the Spanish government does not allow researchers to share individual participant data.

REFERENCES:
- [Background] Ahles TA. Brain vulnerability to chemotherapy toxicities. Psychooncology. 2012 Nov;21(11):1141-8. doi: 10.1002/pon.3196. Epub 2012 Oct 1. PMID 23023994
- [Background] Asher A, Myers JS. The effect of cancer treatment on cognitive function. Clin Adv Hematol Oncol. 2015 Jul;13(7):441-50. PMID 26353040
- [Background] Boykoff N, Moieni M, Subramanian SK. Confronting chemobrain: an in-depth look at survivors' reports of impact on work, social networks, and health care response. J Cancer Surviv. 2009 Dec;3(4):223-32. doi: 10.1007/s11764-009-0098-x. Epub 2009 Sep 16. PMID 19760150
- [Background] Bray VJ, Dhillon HM, Bell ML, Kabourakis M, Fiero MH, Yip D, Boyle F, Price MA, Vardy JL. Evaluation of a Web-Based Cognitive Rehabilitation Program in Cancer Survivors Reporting Cognitive Symptoms After Chemotherapy. J Clin Oncol. 2017 Jan 10;35(2):217-225. doi: 10.1200/JCO.2016.67.8201. Epub 2016 Oct 28. PMID 28056205
- [Background] Pendergrass JC, Targum SD, Harrison JE. Cognitive Impairment Associated with Cancer: A Brief Review. Innov Clin Neurosci. 2018 Feb 1;15(1-2):36-44. PMID 29497579
- [Background] Fernandes HA, Richard NM, Edelstein K. Cognitive rehabilitation for cancer-related cognitive dysfunction: a systematic review. Support Care Cancer. 2019 Sep;27(9):3253-3279. doi: 10.1007/s00520-019-04866-2. Epub 2019 May 30. PMID 31147780
- [Background] Hardy SJ, Krull KR, Wefel JS, Janelsins M. Cognitive Changes in Cancer Survivors. Am Soc Clin Oncol Educ Book. 2018 May 23;38:795-806. doi: 10.1200/EDBK_201179. PMID 30231372
- [Background] Hutchinson AD, Hosking JR, Kichenadasse G, Mattiske JK, Wilson C. Objective and subjective cognitive impairment following chemotherapy for cancer: a systematic review. Cancer Treat Rev. 2012 Nov;38(7):926-34. doi: 10.1016/j.ctrv.2012.05.002. Epub 2012 Jun 2. PMID 22658913
- [Background] Janelsins MC, Heckler CE, Peppone LJ, Kamen C, Mustian KM, Mohile SG, Magnuson A, Kleckner IR, Guido JJ, Young KL, Conlin AK, Weiselberg LR, Mitchell JW, Ambrosone CA, Ahles TA, Morrow GR. Cognitive Complaints in Survivors of Breast Cancer After Chemotherapy Compared With Age-Matched Controls: An Analysis From a Nationwide, Multicenter, Prospective Longitudinal Study. J Clin Oncol. 2017 Feb 10;35(5):506-514. doi: 10.1200/JCO.2016.68.5826. Epub 2016 Dec 28. PMID 28029304
- [Background] Bail J, Meneses K. Computer-Based Cognitive Training for Chemotherapy-Related Cognitive Impairment in Breast Cancer Survivors. Clin J Oncol Nurs. 2016 Oct 1;20(5):504-9. doi: 10.1188/16.CJON.504-509. PMID 27668370
- [Background] Van Dyk K, Bower JE, Crespi CM, Petersen L, Ganz PA. Cognitive function following breast cancer treatment and associations with concurrent symptoms. NPJ Breast Cancer. 2018 Aug 17;4:25. doi: 10.1038/s41523-018-0076-4. eCollection 2018. PMID 30131974
- [Background] Von Ah D, Habermann B, Carpenter JS, Schneider BL. Impact of perceived cognitive impairment in breast cancer survivors. Eur J Oncol Nurs. 2013 Apr;17(2):236-41. doi: 10.1016/j.ejon.2012.06.002. Epub 2012 Aug 14. PMID 22901546
- [Background] Zeng Y, Dong J, Huang M, Zhang JE, Zhang X, Xie M, Wefel JS. Nonpharmacological interventions for cancer-related cognitive impairment in adult cancer patients: A network meta-analysis. Int J Nurs Stud. 2020 Apr;104:103514. doi: 10.1016/j.ijnurstu.2019.103514. Epub 2020 Jan 3. PMID 32004776